CLINICAL TRIAL: NCT04438109
Title: Clinical Outcome of the Dynamic Reconstruction of the Medial Patellofemoral Ligament (MPFL) - a Retrospective Case Series
Brief Title: Clinical Outcome of the Dynamic Reconstruction of the Medial Patellofemoral Ligament (MPFL)
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 8262_BO_K_2019
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Patellar Luxation; Patellar Instability
Keywords: knee; MPFL reconstruction; patella instability; patella dislocation
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a single surgical center, 213 consecutive patients with 221 knees were surgically treated for recurrent lateral patellar dislocation between 07/2010 and 12/2016. All patients obtained dynamic reconstruction of the MPFL with detachment of the gracilis tendon at the pes anserinus while maintaining the proximal origin at the gracilis muscle. Patellar fixation was performed by oblique transpatellar tunnel transfer and tenodesis screw. Follow-up data including Kujala-, BANFF- and Norwich patellar instability score as well as Return-to-Sport and pain level were collected at a minimum follow-up of 2 years

DETAILED DESCRIPTION:
Patients were identified through the hospitals database using OPS-Codes for MPFL reconstruction. The included surgeries were performed from 07/2010 to 12/2016 in a single orthopedic hospital.

Inclusion criteria:

* Dynamic MPFL-reconstruction (primary and revision surgery) including cartilage procedure
* Age of 18 years or older at a minimum of 24 months follow up

Exclusion criteria:

* Diagnosis of connective tissue disease
* Neurological diseases including patella associated spasticity and
* Concomitant alignment correction surgery including femoral/tibial osteotomy, trochleoplasty and tibial tubercle transfer

  213 Patients with 221 knees (8 bilateral) met the inclusion criteria. All patients were contacted by mail or phone to independently answer questionnaires.

Surgical technique:

The technique was performed according to the description by Ostermeier et al.. Briefly, the gracilis tendon is detached at its insertion site at the pes anserinus after opening the sartorius fascia. Instead of transferring the tendon through a subligamentous tunnel of the medial collateral ligament, as detailed in the original description of the technique, the tendon was passed around the incised sartorius fascia. From around the sartorius fascia the gracilis tendon is shuttled subcutaneously to the medial patellar margin, allowing the sartorius fascia to act as a pulley for the transferred tendon. Due to the dynamic reconstruction technique, the course of the graft appears to be more oblique compared to the static technique with femoral fixation at Schöttle's point. Fixation of the tendon is achieved by passing it through a transpatellar drill hole extending from the proximal medial patellar margin to the lateral patellar margin. The tendon is then tensioned with the knee in 30 degrees of flexion and fixed with a bioabsorbable tenodesis screw.

Data collection was performed by self-administered questionnaires, which were sent to the patients.

The medical records and radiographs of all patients were reviewed for demographic information (age, sex) and to identify complications related to the surgical procedure. Complications were categorized as major if the patient returned to the operating room or required hospitalization after the index procedure. Complications were categorized as minor complications if they were treated on an outpatient basis.

Rating of the results was performed using the Kujala score, the Norwich Patellar Instability Score and the BANFF Score.

Pain level was recorded using the visual analogue scale (VAS, 0 = no pain, 10 = severe pain). General satisfaction with treatment outcomes was evaluated by questionnaire (1 = excellent, 2 = very good, 3 = good, 4 = fair, 5 = poor, 6 = very poor) and by asking patients whether they would undergo the procedure again. Furthermore, information on patient characteristics, recurrence of dislocation, revision surgery, and other postoperative complications were recorded.

Postoperative x-rays were analyzed concerning intraoperative complications (e.g. fractures or patellar drill hole malpositioning).

ELIGIBILITY:
Inclusion Criteria:

* Patients with MPFL reconstruction and possible accompanying interventions
* Age >18 years

Exclusion Criteria:

* Known hereditary connective tissue diseases (e.g. Ehlers-Danlos syndrome)
* Known neurogenic diseases
* Significant further musculoskeletal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were identified through the hospitals database using OPS-Codes for MPFL reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2021-02-27 (Actual)

PRIMARY OUTCOMES:
Kujala score | 24 months postoperative
  The Kujala Anterior Knee Pain Scale is a patient reported assessment of patellofemoral disorders that assesses subjective symptoms and functional limitations.
  The score consists of 13 questions that add up to a total of 100 points. Minimum: 0 (worst), Maximum: 100 (best)
Norwich Patellar Instability Score (NPI Score) | 24 months postoperative
  The Norwich Patellar Instability Score is a patient reported assessment of patellofemoral instability.
  The score consists of 19 questions with a special weighting for every question. The results are presented in percent. Range: 0% (best) to 100% (worst)
BANFF Score | 24 months postoperative
  The Banff Score is a patient reported assessment of patellofemoral disorders that assesses patella instability.
  The score consists of 23 questions. Minimum: 0 (worst), Maximum: 100 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopädische Klinik der Medizinischen Hochschule Hannover im DIAKOVERE Annastift, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Horstmann H, Karkosch R, Berg A, Becher C, Petri M, Smith T. The novel dynamic MPFL-reconstruction technique: cheaper and better? Arch Orthop Trauma Surg. 2022 Aug;142(8):2011-2017. doi: 10.1007/s00402-021-04198-z. Epub 2021 Oct 11. PMID 34633513